CLINICAL TRIAL: NCT06845189
Title: Role of Modified Robbery Exercises on Scapular Dyskinesis in Patients With Frozen Shoulder
Brief Title: Role of Modified Robbery Exercises on Scapular Dyskinesis in Frozen Shoulder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CMH Lahore Medical College and Institute of Dentistry (Other)
Collaborators: University of Lahore (Other)
Responsible Party: Principal Investigator, Wajida Perveen, Associate Professor & HOD DPT, CMH Lahore Medical College and Institute of Dentistry
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 109/ERC/CMH/LMC
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Frozen Shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Robbery Exercises Group (Experimental): the participants will receive prescribed set of Modified Robbery exercises
  Interventions: Other: Modified Robbery Exercises
- Conventional Physiotherapy treatment (Active Comparator): the participants will receive conventional physiotherapy treatment for Frozen shoulder.
  Interventions: Other: Conventional Physiotherapy Treatment

INTERVENTIONS:
Other: Modified Robbery Exercises — Prescribed set of Modified Robbery exercises will be applied
  Arms: Modified Robbery Exercises Group
Other: Conventional Physiotherapy Treatment — Conventional Physiotherapy Treatment for Frozen Shoulder
  Arms: Conventional Physiotherapy treatment

SUMMARY:
The study aims to find out the role of the modified robbery exercises in the management of scapular dyskinesia in patients with frozen shoulders. This single-blind randomized clinical study will be conducted at approved study center in Lahore Pakistan in line with the ethical principles stated in Declaration of Helsinki. Pain, muscle Activation, ROM, scapular dyskinesia, muscle strength, functional limitation and participants' wellbeing will be recorded at baseline, after week three, and after week six in both intervention and control groups.

DETAILED DESCRIPTION:
Scapular Dyskinesia is regarded as the altered scapular kinematics, presenting with increased scapular upward rotation and eminence of the medial border in patients with shoulder injuries. Patients with frozen shoulder present with a certain degree of scapular dyskinesia. The objective of the study is to find out the role of the modified robbery exercises in the management of scapular dyskinesia in patients with frozen shoulders. This single-blind randomized clinical study will be conducted at approved study center in Lahore Pakistan. The study will abide by the ethical principles in line with the Declaration of Helsinki. Baseline data of the participants of pain, muscle Activation, ROM, scapular dyskinesia, muscle strength, functional limitation and participants' wellbeing will be recorded. Group A will receive the modified robbery exercises three days a week for six weeks, group B will receive the conventional physical therapy protocol three days a week for six weeks. Outcomes will be assessed at baseline, after week three, and after week six.

Data will be recorded using questionnaires, proforma and the other listed outcome measurement tools. on the base of normality of the data appropriate parametric test or non-parametric test will be applied for intra and inter group comparison.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders
* Patients of age 35 to 55 years
* Modified Lateral Scapular Slide Test score > 1.4 cm
* Pain on VAS ≥4 out of 10.
* Pain in the shoulder for at least 3 months
* Diagnosed unilateral frozen shoulder
* Limited Scapular upward rotation, Capsular pattern (more limited external rotation than abduction),
* Scapular dispositioning and visible Inferior medial border prominence.

Exclusion Criteria:

* Patients with frozen shoulders having less than 90 degrees of flexion and abduction.
* Participants with cervical radicular pain
* Pregnant females
* Presence of red flags to the treatment
* History of recent trauma to the spine or the shoulder complex.
* History of recent shoulder surgery
* Any neurological deficit i.e winged scapula
* Other pathologies like cervical myelopathy and prolapsed cervical disc.
* Known cases of neurological, radiculopathy, and inflammatory diseases.
* Having spinal deformities such as scoliosis or kyphosis.
* Vestibular or respiratory disorder, Auditory or cognitive impairment
* Taking medication that may affect the balance and coordination.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2026-01-25 (Actual); Study Completion 2026-08-25 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | baseline, at week 3 and at week 6
  Pain intensity will be measured using Visual Analogue Scale.
Scapular Dyskinesia | baseline, at week 3 and at week 6
  Score of Modified Lateral Scapular Slide Test using Vernier caliper
Range of scapular and shoulder Motion | baseline, at week 3 and at week 6
  Range of Motion of selected movements will be measured on Goniometer
Muscle Strength | baseline, at week 3 and at week 6
  Muscle Strength of selected muscles will be measured by manual muscle testing
Muscle activation | baseline, at week 3 and at week 6
  Muscle activation of selected muscles will be measured by Electromyography Biofeedback

SECONDARY OUTCOMES:
shoulder functions | baseline, at week 3 and at week 6
  shoulder functions will be assessed using Shoulder pain and disability Index (SPADI-U)
Well-being | baseline, at week 3 and at week 6
  Well-being of the participants will be assessed using the WHO 5 Wellbeing Index

CONTACTS AND LOCATIONS:
Overall Officials: Wajida Perveen, Principal Investigator — School of Allied Health Sciences, CMH Lahore Medical College & IOD (NUMS Rawalpindi)
Locations (1):
- School of Allied Health Sciences, CMH Lahore Medical College & Institute of Dentistry, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No